CLINICAL TRIAL: NCT00961454
Title: A Pilot Study to Evaluate the Ability of Photobiomodulation to Alter Cerebral Blood Flow in the Frontal Poles and to Affect the Emotional Status of Patients With Major Depression
Brief Title: Photobiomodulation to Alter Cerebral Blood Flow and to Affect the Emotional Status of Patients With Major Depression
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Responsible Party: Michael Hamblin, Massachusetts General Hospital
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2008P-000937
Record Dates: First submitted 2009-08-18; First posted 2009-08-19 (Estimated); Last update posted 2009-08-19 (Estimated); Status verified 2009-08

CONDITIONS: Major Depression; Anxiety Disorder; Post-Traumatic Stress Disorder; Substance Abuse Disorder
Keywords: Major depressive disorder, anxiety disorders, treatments, photobiomodulation, near infra-red phototherapy, cerebral blood flow
MeSH Terms: conditions — Depressive Disorder, Major; Anxiety Disorders; Stress Disorders, Post-Traumatic; Substance-Related Disorders | interventions — Low-Level Light Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Device: Photobiomodulation with a super-luminous light emitting diode — The treatment will consist of applying PBM in the form of a super-luminous LED with an output of 250 mW/cm2 at a wavelength of 815 nm with a full width half maximum of 40 nm when applied at 4 mm from the skin. The treatment will consist of the exposure to the light for 4 minutes (total delivered fluence per spot of 60 J/cm2) at each of 4 sites on the forehead that correspond to the 10-20 EEG sites, F3, and F4.
  Other Names: Near infra-red light

SUMMARY:
A pilot study to evaluate the ability of photobiomodulation to alter cerebral blood flow in the frontal poles and to affect the emotional status of patients with major depression.

DETAILED DESCRIPTION:
We wish to study whether photobiomodulation (PBM) with near infrared (NIR) light emitting diodes (LED), a non-ionizing phototherapy, in patients with major depression, can acutely alter frontal brain blood flow measured by near infrared spectroscopy (NIRS).

Secondarily, we will examine whether PBM can improve emotional state immediately and over the following month.

We see this as a pilot study to gather preliminary data that will guide future studies.

ELIGIBILITY:
Inclusion Criteria:

* All patients must be right handed, between the ages of 18 and 60, and meet criterion for depression on a Structured Clinical Diagnostic Interview
* Enrollment will be made without regard to gender or ethnicity
* Patients who are receiving treatment for depression, either psychological or pharmacological, may continue their treatment during the time of the study, but will be asked to try not to alter their treatment from one month prior to the onset of the experiment until its conclusion. If they must alter their treatment, the patient will continue in the study for observation, but will be excluded from any follow-up statistical comparisons

Exclusion Criteria:

* Past history of psychotic disorder (including schizophrenia or schizoaffective disorder
* Bipolar disorder
* Obsessive compulsive disorder)
* Substance abuse disorder that has been active with the past 6 months,
* A history of violent behavior
* A history of a past suicide gesture or attempt
* A history of current suicidal ideation
* A history of a neurological condition (e.g. epilepsy, traumatic brain injury, stroke)
* Pregnancy
* Current acute or chronic medical condition requiring a medications that has psychological side-effects
* Any person whom we judge to have an impaired decision-making capacity

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 10 (Actual)
Dates: Start 2009-01; Primary Completion 2009-06 (Actual); Study Completion 2009-06 (Actual)

PRIMARY OUTCOMES:
Hamilton Depression Rating Scale | Before treatment (baseline), 2-weeks after treatment, and 4-weeks after treatment

SECONDARY OUTCOMES:
Hamilton Anxiety Rating Scale | Before treatment, 2-weeks after treatment, and 4-weeks after treatment
Hamilton Anxiety Rating Scale | Before treatment (baseline), 2-weeks after treatment, and 4-weeks after treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Fredric - Schiffer, M.D., Study Director — McLean Hospital and the Harvard Medical School; Robert H Webb, Ph.D., Study Chair — Massachusetts General Hospital; Andrea Johnston, BA, Study Chair — Massachusetts General Hospital; Martin H Teicher, M.D., Ph.D., Study Chair — Mclean Hospital
Locations (1):
- Wellman Center for Photomedicine, Massachusetts General Hospital, Boston, Massachusetts, United States

REFERENCES:
- [Derived] Schiffer F, Johnston AL, Ravichandran C, Polcari A, Teicher MH, Webb RH, Hamblin MR. Psychological benefits 2 and 4 weeks after a single treatment with near infrared light to the forehead: a pilot study of 10 patients with major depression and anxiety. Behav Brain Funct. 2009 Dec 8;5:46. doi: 10.1186/1744-9081-5-46. PMID 19995444